CLINICAL TRIAL: NCT01112995
Title: A Pilot Randomized Trial to Determine the Efficacy of a Probiotic, Lactobacillus Rhamnosus for Reducing Colonization by Methicillin-resistant Staphylococcus Aureus (MRSA)
Brief Title: A Pilot Trial to Determine the Efficacy of Lactobacillus Rhamnosus for Reducing Colonization by Methicillin-resistant Staphylococcus Aureus (MRSA) (PROSE)
Acronym: PROSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008-0023
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-04

CONDITIONS: Infection
Keywords: Probiotic; Lactobacillus; Antibiotic resistance
MeSH Terms: conditions — Infections | interventions — Sugars; trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): subjects will be given a pill formulation of a probiotic Lactobacillus rhamnosus to be taken once a day.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus
- Sugar pill (Placebo Comparator): placebo identical to the active product will be given
  Interventions: Dietary Supplement: Sugar pill (placebo)

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus — 1 pill formulation to be given once a day for 4 weeks
  Other Names: Yoplait; Activia
  Arms: Probiotic
Dietary Supplement: Sugar pill (placebo) — placebo identical to the active product will be given
  Other Names: splenda
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to investigate the feasibility, safety and efficacy of oral probiotic, Lactobacillus rhamnosus versus oral placebo for reducing colonization by MRSA.

DETAILED DESCRIPTION:
Healthcare-associated infections are an important threat to patient safety. Currently, between 5 and 10 percent of patients admitted to acute care hospitals acquire one or more infections; healthcare-associated infections affect approximately 2 million patients each year in the United States, result in 90,000 deaths, and are associated with an added cost of $4.5 to $5.7 billion per year. Seventy percent of healthcare-associated infections are caused by antimicrobial resistant bacteria, such as methicillin-resistant Staphylococcus aureus (MRSA), resulting in increased antimicrobial usage, morbidity and mortality, making prevention of multiresistant bacteria essential.

Eradication of colonization has been shown to greatly reduce infection; however, there are no reliable means of providing sustained eradication of colonization. No effective means of eradicating MRSA colonization exist.

Probiotics containing strains of lactobacilli represent a novel approach to the prevention and control of antimicrobial resistance and have been studied extensively for a variety of infections. Even though various studies have shown probiotics to be effective for prevention of vaginal infections, urinary tract infections, etc no studies have examined the potential of probiotics to eradicate colonization by resistant pathogens, such as MRSA.

ELIGIBILITY:
Inclusion Criteria:

* subjects will be male or female
* 18 years of age or older
* may or may not be hospitalized
* able to take oral medications
* have been found to be colonized with MRSA or at high risk of being colonized by MRSA and are not taking antibiotics

Exclusion Criteria:

* people on antibiotics will not be eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The main outcomes will be the proportion of patients colonized with MRSA at 4 weeks, 8 weeks, 12 weeks and 24 weeks following start of treatment. | 24 weeks

SECONDARY OUTCOMES:
Incidence of clinical infections will be assessed in the one year following enrollment into the study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD, Ph.D, Principal Investigator — University of Wisconsin Department of Medicine (Infectious Disease)
Locations (1):
- University of Wisconsin Hospital, Madison, Wisconsin, United States